CLINICAL TRIAL: NCT05051397
Title: Evaluation of the Effect of Moderate and Controlled Hypercapnia on Ischemic Penumbra Vascular Collaterality During General Anesthesia for Anterior Circulation Acute Ischemic Stroke Mechanical Thrombectomy
Brief Title: CO2 Modulation in Endovascular Thrombectomy for Acute Ischemic Stroke
Acronym: COMET-AIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COMET-AIS (AOI 2020 Chabanne); AOI... (Other Grant/Funding Number: CHU Clermont-Ferrand)
Record Dates: First submitted 2021-07-09; First posted 2021-09-21 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke, Acute; Thrombectomy; Anesthesia, General; Cerebrovascular Circulation; Carbon Dioxide
Keywords: mechanical thrombectomy; large vessel occlusion stroke; carbon dioxide tension; cerebral blood flow; general anesthesia; cerebral collateral circulation
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HYPERCAPNIA (Experimental): Under general anesthesia with mechanical ventilation, PaCO2=50mmHg will be targeted
  Interventions: Biological: HYPERCAPNIA
- NORMOCAPNIA (Active Comparator): Under general anesthesia with mechanical ventilation, PaCO2=40mmHg will be targeted
  Interventions: Biological: NORMOCAPNIA

INTERVENTIONS:
Biological: HYPERCAPNIA — Controlled moderate hypercapnia PaCO2 50mmHg under general anesthesia with mechanical ventilation
  Arms: HYPERCAPNIA
Biological: NORMOCAPNIA — Controlled normocapnia PaCO2 40mmHg under general anesthesia with mechanical ventilation
  Arms: NORMOCAPNIA

SUMMARY:
Acute ischemic stroke due to large vessel occlusion is responsible of cerebral blood flow impairment with a progressive and extensive ischemic process. Cerebral collateral circulation may preserve an ischemic penumbra that could recover providing timely reperfusion of the occluded vessel. Mechanical thrombectomy is the standard of care for anterior circulation large vessel reperfusion. Strategy to promote cerebral blood flow in collateral circulation before reperfusion is scarce and rely mainly on blood pressure maintenance. Carbon dioxide is a potent cerebral vasodilator that could enhance collateral circulation blood flow and cerebral protection before reperfusion. General anesthesia with endotracheal mechanical ventilation could be used for thrombectomy and give the opportunity to modulate and control carbon dioxide tension in the blood. This study will test the effect of moderate hypercapnia on penumbral collateral circulation before reperfusion during mechanical thrombectomy for anterior circulation acute ischemic stroke under general anesthesia.

DETAILED DESCRIPTION:
Study will compare 2 groups of patients treated for anterior circulation large vessel occlusion stroke thrombectomy under general anesthesia.

After anesthetic evaluation, patients will be randomized to receive moderate hypercapnia targeting an arterial CO2 tension (PaCO2) of 50mmHg or normocapnia targeting a PaCO2 of 40mmHg.

The anesthetic protocol will use:

* Rapid sequence induction for orotracheal intubation with PROPOFOL 2mg/Kg and SUXAMETHONIUM 1mg/Kg
* SUFENTANIL 0,1 µg/Kg and CISATRACURIUM 0,1mg/Kg
* Maintenance with intravenous continuous infusion of PROPOFOL targeting a BISpectral index 40 to 60
* Systolic blood pressure will have to be maintained +/- 10% of preoperative baseline value with limits between 120 and 185mmHg (with NOREPINEPHRINE as needed)
* Mechanical ventilation will use Tidal Volume of 7mL/Kg of ideal body weight, respiratory rate of 15/minute, End expiratory pressure of 5cmH2O. FiO2 will target SpO2 95-98%. Initial End Tidal CO2 (EtCO2) target will be 35mmHg.
* A first arterial blood gas analysis at groin puncture will evaluate CO2 alveolar-arterial gradient in order to obtain the expected PaCO2 in each group with respiratory rate modulation on the ventilator.
* ASITN baseline collaterality score will be evaluated at initial angiography with normocapnia in each group. A second evaluation of ASITN will be done just before deployment of intraarterial revascularisation device in hypercapnia or normocapnia depending on randomisation group.
* Targeted PaCO2 will have to be maintained using EtCO2 surrogate until the end of procedure.
* A second arterial blood gas analysis at the end of procedure will evaluate final PaCO2.

ELIGIBILITY:
Inclusion Criteria:

• Large vessel occlusion anterior circulation stroke (terminal carotid artery and/or middle cerebral artery M1-M2 segment) eligible to mechanical thrombectomy under general anesthesia

Exclusion Criteria :

* Active smoker
* Chronic respiratory failure with ambulatory oxygen supplementation
* Obesity with BMI>40Kg/ m2
* Intubation before the procedure
* Heart failure with intolerance to decubitus
* Severe renal failure
* Suspected elevated intracranial pressure
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-07-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
ASITN cerebral vascular collaterality score > 2 | Before reperfusion of the occluded vessel
  American Society of Interventional and Therapeutic Neuroradiology (ASITN) cerebral vascular collaterality score ranges from 0 (no collaterals visible to the ischemic site) to 4 (complete and rapid collateral blood flow to the vascular bed in the entire ischemic territory by retrograde perfusion). A score > 2 indicate at least collaterals with slow but complete angiographic blood flow of the ischemic bed by the late venous phase.

SECONDARY OUTCOMES:
ASITN cerebral vascular collaterality score | • At initial angiography in normocapnia and • Before reperfusion at randomized arterial CO2 tension level
  American Society of Interventional and Therapeutic Neuroradiology (ASITN) variation during the procedure
Volume of cerebral infarction | 24 hours after stroke
  Evaluated with Magnetic Resonance Imaging in milliliters
Progression of cerebral infarction | 24 hours after stroke
  Evaluated with Magnetic Resonance Imaging or Computed Tomography in milliliters depending on type of radiological modality for patient selection
Neurological clinical outcome | 3 months
  Ordinal and dichotomized modified rankin scale (mRS) ranging from 0 (no disability) to 6 (death); good outcome will be defined as mRS 0-2.

OTHER OUTCOMES:
Pial Vascular Collaterality within the symptomatic ischemic territory at admission | At admission
  Pial Vascular collaterality evaluated at admission with CT or MRI during patient selection for thrombectomy using the Pial Arterial Filling Score (from 0 indicated no collaterality to 5 indicating excellent collaterality)
Arterial carbon dioxide tension | At groin puncture and at the end of procedure
  Arterial carbon dioxide tension will be measured at 2 time points.
Cerebral infarction extension | Before thrombectomy and at day 1
  The Alberta Stroke Program Early Computed Tomography Score (ASPECTS) is an imaging measure of the extent of ischemic stroke. Scores range from 0 to 10, with higher scores indicating a smaller infarct core.
Reperfusion assessed by mTICI | End of procedure
  The modified Treatment In Cerebral Ischemia (mTICI) reperfusion scale ranging from 0 (no perfusion) to 3 (full perfusion with filling of all distal Branches). Good reperfusion will be defined as a score of 2B-3.
Procedural delay | End of procedure
  Time frame from angiosuite admission to groin puncture to reperfusion if any
Number of procedural anesthetic and radiological complications | End of procedure
  Procedural Safety outcomes
Number of Death and neurological complications | Day 7
  Safety outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Russell Chabanne, MD MSc, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schonenberger S, Henden PL, Simonsen CZ, Uhlmann L, Klose C, Pfaff JAR, Yoo AJ, Sorensen LH, Ringleb PA, Wick W, Kieser M, Mohlenbruch MA, Rasmussen M, Rentzos A, Bosel J. Association of General Anesthesia vs Procedural Sedation With Functional Outcome Among Patients With Acute Ischemic Stroke Undergoing Thrombectomy: A Systematic Review and Meta-analysis. JAMA. 2019 Oct 1;322(13):1283-1293. doi: 10.1001/jama.2019.11455. PMID 31573636
- [Background] Slupe AM, Kirsch JR. Effects of anesthesia on cerebral blood flow, metabolism, and neuroprotection. J Cereb Blood Flow Metab. 2018 Dec;38(12):2192-2208. doi: 10.1177/0271678X18789273. Epub 2018 Jul 16. PMID 30009645
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Background] Willie CK, Macleod DB, Shaw AD, Smith KJ, Tzeng YC, Eves ND, Ikeda K, Graham J, Lewis NC, Day TA, Ainslie PN. Regional brain blood flow in man during acute changes in arterial blood gases. J Physiol. 2012 Jul 15;590(14):3261-75. doi: 10.1113/jphysiol.2012.228551. Epub 2012 Apr 10. PMID 22495584
- [Background] Olsen TS, Larsen B, Herning M, Skriver EB, Lassen NA. Blood flow and vascular reactivity in collaterally perfused brain tissue. Evidence of an ischemic penumbra in patients with acute stroke. Stroke. 1983 May-Jun;14(3):332-41. doi: 10.1161/01.str.14.3.332. PMID 6658900